CLINICAL TRIAL: NCT07093593
Title: Emergence of Bacterial Resistance to Antibiotics in the Digestive Microbiota of Patients Treated With Anticancer Drugs (Clinical Component of the RAMA Project)
Brief Title: Emergence of Bacterial Resistance to Antibiotics in the Digestive Microbiota of Patients Treated With Anticancer Drugs
Acronym: RAMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025-A00013-46
Record Dates: First submitted 2025-06-02; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancers; Endometrial Cancer; Gynecological Cancers; Pancreatic Adenocarcinoma; Upper Aerodigestive Tract Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — Blood Specimen Collection; Receptors, Lymphocyte Homing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All cohorts (Experimental): For each cohort :
  * Collect of stool samples (cycle 1 and cycle 3)
  * Collect of blood samples (5 x 6 mL EDTA tubes) => Cycle 1 and Cycle 3
  Interventions: Other: Mandatory biological samples (blood and sell)

INTERVENTIONS:
Other: Mandatory biological samples (blood and sell) — At cycle 1 and Cycle 3 :
  * Stool sample collection
  * Blood sample collection (5 EDTA tubes)

SUMMARY:
Solid cancers are frequently treated with chemotherapies that target the DNA of cancer cells. It has recently come to light that bacteria are also the target of chemotherapies used in oncology. The results of current studies demonstrate the close link between the composition of the microbiota, the immune system, toxicity and the efficacy or otherwise of anti-cancer treatments.

In this context, the study will measure the influence of treatment with anticancer molecules known to activate the bacterial SOS response on the emergence of antibiotic-resistant commensal bacteria in the gut microbiota of cancer patients. Furthermore, this study will investigate the existence of a close link between changes in the intestinal microbiota determined by the induction or non-induction of the SOS response, bacterial translocation, the integrity of the intestinal barrier and the antitumor immune response.

The RAMA trial plans to collect stool and blood samples from two different cohorts of patients:

* Unexposed cohort: patients receiving anti-cancer treatment that does not induce bacterial SOS response.
* Exposed cohort: patients receiving anti-cancer treatment inducing the bacterial SOS response.

Patients' stools will be collected within 7 days of their first chemotherapy treatment and within 7 days of the 3rd chemotherapy cycle. Two blood samples will be taken at the same time as the stool samples.

The results obtained from this prospective clinical research will then be investigated in two experimental laboratory models.

The aim is to demonstrate that cytotoxic anticancer drugs promote the emergence of antibiotic-resistant commensal bacteria, by means of this large-scale study comprising a clinical component, which is the subject of the research presented in this protocol, combined with laboratory research components.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18
* Chemotherapy-naive patients.
* Patients due to start chemotherapy/radio chemotherapy who meet the criteria of the cohorts listed below :

  1. Squamous cell carcinoma of the upper aerodigestive tract (Non-metastatic, locally advanced, operable or not; Patients receiving concomitant radiochemotherapy using a platinum salt (cisplatin, carboplatin))
  2. Cervical and endometrial cancer (ocally advanced, Non-metastatic; Patients receiving concomitant radiochemotherapy using a platinum salt (cisplatin, carboplatin))
  3. Gynecological cancer (advanced stage ; Patient to receive platinum salt + paclitaxel chemotherapy)
  4. Mammary carcinoma (localised; Patient to receive adjuvant or neoadjuvant chemotherapy with epirubicin and cyclophosphamide without other associated treatment (targeted therapy / immunotherapy))
  5. Urothelial carcinoma (all stage ; Patient to receive neoadjuvant or adjuvant chemotherapy with platinum salt and gemcitabine)
  6. Pancreatic adenocarcinoma (localised or metastatic ; Patients to be treated with gemcitamine alone or in combination with nab-paclitaxel)
* OMS ≤ 2
* Affiliation with a French social security scheme or beneficiary of such a scheme.
* Signed informed consent indicating that the patient has understood the purpose and procedures of the study and agrees to participate in the study and to abide by the study requirements and restrictions

Exclusion Criteria:

* Patients unable to collect / send stools for medical, geographical, social or psychological reasons.
* Patients who have already received chemotherapy/radiochemotherapy.
* Use of anti-infectives for systemic use within 6 months prior to the first sampling, or any other concomitant disease/condition that may influence stool analysis.
* Pregnant women and nursing mothers.
* Persons deprived of their liberty by judicial or administrative decision; persons under compulsory psychiatric care; persons admitted to a health or social institution for purposes other than research.
* Adults subject to a legal protection measure - safeguard of justice, guardianship or curatorship - or unable to express their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2032-09-01 (Estimated); Study Completion 2032-09-01 (Estimated)

PRIMARY OUTCOMES:
Determine whether the digestive microbiota of patients exposed to SOS-inducing cytotoxic cancer drugs favors the emergence of antibiotic-resistant commensal bacteria compared to patients exposed to other non-SOS-inducing cytotoxic cancer drugs. | up to 3 months
  The primary endpoint is the emergence of antibiotic-resistant Enterobacteriaceae, defined as the presence of Enterobacteriaceae resistant to 3rd-generation cephalosporins and/or fluoroquinolones on the sample taken within 7 days of administration of the 3rd cycle of chemotherapy, compared with the pretreatment initiation sample taken within 7 days of administration of the first cycle of chemotherapy.

IPD SHARING:
Plan to Share IPD: No